CLINICAL TRIAL: NCT01740830
Title: The Effect of Anodal tDCS on Motor Learning in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Koen Cuypers, Drs. Koen Cuypers, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MECU2012-003
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Anodal tDCS; Recruitment Curves
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anodal tDCS (Active Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS) (Neuroconn DC-stimulator)
- Sham tDCS (Sham Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS) (Neuroconn DC-stimulator)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) (Neuroconn DC-stimulator) — The anode will be fixed over the primary motor cortex. The cathode will be fixed over the contralateral supraorbital region.
  Other Names: Neuroconn DC-stimulator

SUMMARY:
The current study investigates the effects of tDCS in patients with multiple sclerosis (MS). The investigators hypothesize that anodal tDCS will increase motor performance in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* male and female

Exclusion Criteria:

* relapse in the last 3 months
* when not suitable for tDCS (screening)
* if TMS measures can not be completed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Motor performance on a unimanual sequence learning task | Baseline, during training and POST (30 min after baseline) intervention
  Patients were instructed to perform a unimanual sequence-learning task consisting of sequential finger presses. The following parameters were measured: Correct sequences/mean inter tap interval (ITI), percentage correct key presses/mean ITI, percentage correct sequences, percentage correct key presses, mean ITI, and mean correct sequences in the performance interval.